CLINICAL TRIAL: NCT04528368
Title: Efficacy and Safety of Using Convalescent Plasma for Treating Patients With COVID-19 Pneumonia Without Indication of Ventilatory Support
Brief Title: Convalescent Plasma for Treating Patients With COVID-19 Pneumonia Without Indication of Ventilatory Support
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: D'Or Institute for Research and Education (Other)
Collaborators: Hospital do Coracao (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 34651120.8.0000.5249
Record Dates: First submitted 2020-08-19; First posted 2020-08-27 (Actual); Last update posted 2021-08-06 (Actual); Status verified 2021-01

CONDITIONS: COVID-19
Keywords: Convalescent plasma; SARS-CoV-2
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Convalescent Plasma + Standard treatment (Experimental): Participants will receive the standard treatment and convalescent plasma
  Interventions: Biological: Convalescent plasma
- Standard treatment (No Intervention): Participants will receive the standard treatment

INTERVENTIONS:
Biological: Convalescent plasma — The intervention group will receive 400 mL of convalescent plasma with a SARS-CoV-2 antispike antibody titer with a dilution ≥ 1: 320.
  Arms: Convalescent Plasma + Standard treatment

SUMMARY:
The COVID-19 pandemic has been spreading continuously, and in Brazil, until August 18, 2020, there have been more than 3,359,000 cases with more than 108,536 deaths, with daily increases. The present study proposes to evaluate the efficacy and safety of using convalescent plasma for treating patients with COVID-19 pneumonia without indication of ventilatory support.

ELIGIBILITY:
Recipient Inclusion Criteria:

* Confirmed diagnosis of COVID-19 by RT-PCR;
* Time between symptom onset and inclusion ≤ 7 days;
* Chest tomography with <50% involvement of the lung parenchyma;
* No indication of ventilatory support at the time of randomization;
* Sign the consent form.

Recipient Exclusion Criteria:

* Contraindication to transfusion or history of previous reactions to blood products for transfusion;
* Pregnant women;
* Limiting comorbidity for administering the therapies provided for in this protocol in the opinion of the investigator.

Donor Inclusion Criteria for Plasmapheresis:

* Convalescent plasma donation will be eligible for patients ≥ 18 years old who had previously confirmed COVID-19 by RT-PCR, which met the criteria adopted by technical notes n13 and 21/2020-CGSH/DAET/SAES/MS;
* SARS-COV-2 negative RT-PCR;
* Asymptomatic for at least 14 days;
* SARS-CoV-2 anti-peak titre with dilution ≥ 1: 320;
* Sign the consent form.

Donor Exclusion Criteria:

* Female gender with previous pregnancy;
* Absence of peripheral venous network compatible with the apheresis procedure;
* Positive or indeterminate result in any of the infectious screening tests;
* Presence of intellectual incapacity to understand the guidelines regarding the risks and benefits of participating in the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-12-11 (Actual); Primary Completion 2021-12-30 (Estimated); Study Completion 2022-01-30 (Estimated)

PRIMARY OUTCOMES:
Area under the curve of SARS-COV-2 viral load obtained from nasopharyngeal and /or oropharyngeal swabs. | 0, 3, 6, 9, 12, 15, 18 and 21 days
  To evaluate the area under the curve of SARSCoV-2 viral load in nasopharyngeal and or oropharyngeal samples on days 0, 3, 6, 9, 12, 15, 18 and 15 after randomization.

SECONDARY OUTCOMES:
Assessment of clinical improvement using an Ordinal Severity Scale | 0, 7, 10, 14, 21 and 28 days
  The seven-point scale is as follows:
  * Death 7 points;
  * Hospital admission for mechanical ventilation plus additional organ support (eg, pressors, RRT, ECMO) = 6 points;
  * Hospital admission for mechanical ventilation = 5 points;
  * Hospital admission for non-invasive ventilation or high-flow oxygen therapy = 4 points;
  * Hospital admission for oxygen therapy (but not requiring high-flow or non-invasive ventilation) = 3 points;
  * Hospital admission but not requiring oxygen therapy = 2 points;
  * Discharged with limitations of activities = 1 point;
  * Discharged with no limitations of activities = 0 point;
Evaluate oxygen saturation | 0, 3, 6, 9, 12, 15, 18 and 21 days
Evaluate oxygen supplementation | 0, 3, 6, 9, 12, 15, 18 and 21 days
Assess respiratory rate | 0, 3, 6, 9, 12, 15, 18 and 21 days
Evaluate the PaO2 / FiO2 ratio (for patients on mechanical mechanisms) | 0, 3, 6, 9, 12, 15, 18 and 21 days
Length of hospital stay | 21 days
Length of stay in intensive care | 21 days
Assess the rate of orotracheal intubation | 21 days
Change in the profile of cytokines/chemokines in both groups | 0, 3, 6, 9, 12, 15, 18 and 21 days
  Quantification by ELISA the levels of 36 molecules determined simultaneously using the Human Cytokine Array Kit da R&D Systems (C5a, IL-4, IL-32 alpha, CD40 ligand, IL-5, CXCL10 / IP-10, G-CSF, IL-6, CXCL11 / I-TAC, GM-CSF, IL-8, CCL2 / MCP-1, CXCL1 / GRO alpha, IL-10, MIF, CCL1 / I-309, IL-12 p70, CCL3 / MIP-1 alpha, ICAM-1, IL-13, CCL4 / MIP-1 beta, IFN -gamma, IL-16, CCL5 / RANTES, IL-1 alpha, IL-17, CXCL12 / SDF-1, IL-1 beta, IL-17E, Serpin E1 / PAI-1, IL-1ra, IL-23, TNF-alpha, IL-2, IL-27 and TREM-1)
Presence of antibodies against SARS-CoV-2 in serum after convalescent plasma administration | 0, 3, 6, 9, 12, 15, 18 and 21 days
Death rate | 7, 10, 14, 21 and 28 days
Rate of transfusion reactions to convalescent plasma infusion | 21 days

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo M Rego, MD, PhD, Principal Investigator — D'Or Institute for Research and Education
Locations (1):
- D'Or Institute for Research and Education, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No